CLINICAL TRIAL: NCT05226533
Title: A Phase 2, Double Blind, Randomized, Placebo Controlled, Multi-center Study to Evaluate the Safety and Efficacy of DWRX2003 in Combination With Remdesivir Following Intramuscular Administration in Moderate-Severe COVID-19 Patients
Brief Title: Clinical Trials to Assess Safety and Efficacy of DWRX2003 Combination With Remdesivir in Moderate to Severe COVID-19 Patients.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped due to difficulties in patient recruitment
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_DWJ1516202
Record Dates: First submitted 2022-02-04; First posted 2022-02-07 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Niclosamide 432mg (Experimental): Niclosamide 432mg (intramuscular injection) + Remdesivir
  Interventions: Drug: DWRX2003
- Niclosamide 960mg (Experimental): Niclosamide 960mg (intramuscular injection) + Remdesivir
  Interventions: Drug: DWRX2003
- Placebo (Placebo Comparator): Placebo (intramuscular injection) + Remdesivir
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DWRX2003 — Intramuscular injection of DWRX2003
  Arms: Niclosamide 432mg; Niclosamide 960mg
Drug: Placebo — Intramuscular injection of placebo
  Arms: Placebo

SUMMARY:
Safety and efficacy of DWRX2003 combination with Remdesivir in moderate to severe COVID-19 patients will be confirmed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of signing the Informed Consent Form (ICF).
* SARS-CoV-2 infection documented by RT-PCR within 7 days prior to randomization.
* Hospitalized patients who meet the criteria of moderate or severe COVID-19.
* Patients who are not pregnant, based on urine pregnancy test during screening, and randomization.
* Female patients of childbearing potential practice effective contraception during the study and be willing and able to continue contraception for 60 days after their dose of study treatment.
* Male patient and/or Female patient's partner agree to use condoms or should have undergone vasectomy or spermicide in addition to female contraception for additional protection against conception for 60 days after their dose of study treatment.
* Patients who are anticipated to available for the entire study period and is capable of understanding and communicating with the investigators and clinical study facility staff.
* Patients who agree to give written informed consent and are willing to participate in the study.

Exclusion Criteria:

* Patients with BMI ≥30 and/or body weight < 40kg
* Patients receiving or who have received antiviral therapy and antiretroviral therapy within 28 days prior to the screening visit.
* Patients who cannot be administered intramuscularly to bilateral ventro-gluteal area.
* Patients with uncontrolled respiratory disease other than COVID-19 pneumonia (i.e. COPD, asthma, cystic fibrosis, etc.)
* Patients who have active malignancy, history of active malignancy or chemotherapy within 1 year from the screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects requiring mechanical ventilation and invasive mechanical ventilation or extra-corporeal membrane oxygenation (ECMO) till day 14. | day 14
  mechanical ventilation and invasive mechanical ventilation or extra-corporeal membrane oxygenation (ECMO) until day 14.

CONTACTS AND LOCATIONS:
Locations (3):
- Indonesia (3):
  - RSUP Fatmawati, Jakarta, DKI Jakarta
  - RSUPN Cipto Mangunkusumo, Jakarta, DKI Jakarta
  - RS. Hasan Sadikin, Bandung, West Java

IPD SHARING:
Plan to Share IPD: No